CLINICAL TRIAL: NCT03692117
Title: Evaluation of Clinical Effectiveness of ECCO2R for the Treatment of Patients With Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Extracorporeal Carbon Dioxide Removal in Severe Chronic Obstructive Pulmonary Disease Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, head of Pulmonary and Critical care medicine ward 4, China-Japan Friendship Hospital
Other Study IDs: 2016YFC1304304-4
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: COPD Exacerbation
Keywords: COPD Exacerbation; Severe; ECCO2R; invasive mechanical ventilation
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Extracorporeal Carbon Dioxide Removal — Place a double lumen catheter in jugular vein, drainage the venous blood in vitro tube, after blood-gas exchange and remove CO2, then return back to the Superior vena cava

SUMMARY:
The conventional treatment for Severe acute exacerbation of Chronic obstructive pulmonary disease including noninvasive respiratory support, invasive respiratory support, etc, but there are many kinds of limitations and complications. Extracorporeal Carbon Dioxide Removal is a life support technology, which can effectively remove CO2. Recently some clinical studies have showed that ECCO2R can effectively improve the AECOPD patient's respiratory failure, avoid intubation and removal of endotracheal intubation. We performed a study to evaluate the clinical effectiveness of ECCO2R in the treatment of AECOPD patients.

DETAILED DESCRIPTION:
With the development of technology, ECCO2R is not difficult to implement in intensive care unit. Many recently clinical studies have showed that ECCO2R can effectively remove CO2, reduce patient breathing work, improve the patient respiratory failure, and avoid endotracheal intubation. But there are also treated failure and high incidence of complications such as bleeding in the AECOPD patients with ECCO2R treatment, and the treatment related to airway management are less mentioned. Therefore, we set a more strict inclusion criteria in AECOPD patients and evaluate the clinical effectiveness and associated risk of ECCO2R in the treatment of AECOPD.

ELIGIBILITY:
Inclusion Criteria:

* NPPV treatment failure:

  1. deterioration or no improvement after treatment with NPPV, pH < 7.25, PaCO2 > 70mmHg
  2. Obvious respiratory distress, RR > 30 times/min
  3. Breathing extreme fatigue

Exclusion Criteria:

* Older than 75 years
* endotracheal intubation or tracheostomy
* obviously a lot of pus yellow phlegm, expectorate difficult
* Chest CT: obviously a wide range of consolidation
* BMI < 20 kg/m2,
* Dysfunction of other organ of extrapulmonary
* serious hemodynamic instability
* severe hypoxemia, PaO2 / FiO2 < 100mmHg
* home noninvasive positive pressure ventilation for a long time
* lung fungal infection
* contraindication of anticoagulation
* Platelet < 80000 per cubic millimeter
* Serum creatinine > 200 umol/L
* cardiac arrest
* Hospice care
* Refused to take part in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with AECOPD accept the NPPV treatment, deterioration or no improvement of Clinical status. we expected them to be avoided endotracheal intubation after treatment with ECCO2R
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
incidence of avoid endotracheal intubation | 30days
  avoid endotracheal intubation and Invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhan, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No